CLINICAL TRIAL: NCT01324193
Title: Effects of Pomegranate Supplementation on Physical Function and Cardiovascular Disease Risk in Chronic Kidney Disease Patients
Brief Title: Pomegranate Supplementation on Physical Function and Cardiovascular Disease Risk in CKD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenneth Wilund (Other)
Responsible Party: Sponsor-Investigator, Kenneth Wilund, Prinicpal Responsible Investigator, University of Illinois at Urbana-Champaign
Organization: University of Illinois at Urbana-Champaign (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10041
Record Dates: First submitted 2011-03-09; First posted 2011-03-28 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Kidney Disease; Cardiovascular Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-diaylsis patients (Other): Chronic Kidney Disease patients not receiving dialysis getting pomegrante Supplementation
  Interventions: Dietary Supplement: Pomegranate extracts
- Dialysis patients (Other): Chronic Kidney Disease patients receiving dialysis getting pomegranate supplementation
  Interventions: Dietary Supplement: Pomegranate extracts

INTERVENTIONS:
Dietary Supplement: Pomegranate extracts — a 1000mg capsule of a purified pomegranate polyphenol supplement (POMx™, POM Wonderful, Inc. Los Angeles, CA)7 days a week for 12 months.

SUMMARY:
Chronic kidney disease (CKD) patients have very low physical function and high rates of cardiovascular disease (CVD) mortality. The objective of the proposed research is to evaluate the effects of dietary supplementation with a pomegranate extract, that contains high amounts of antioxidants, on physical function and CVD risk. Patients with moderate to severe chronic kidney disease that are NOT yet on dialysis tend to have significantly reduced risk factors for cardiovascular disease (and other disorders) compared to dialysis patients. This includes significantly reduced systemic markers of oxidative stress and inflammation. As a result, therapies designed to reduce the risk of CKD co-morbidities may differ significantly in dialysis and pre-dialysis patients. For example, dialysis patients are recommended to INCREASE their intake of dietary protein, while pre-dialysis patients are recommended to DECREASE their protein intake, due to differences in the pathophysiology of the two conditions. The investigators have decided to recruit pre-dialysis patients in addition to dialysis patients in this study because the investigators believe this will help us determine if the efficacy of pomegranate differs between patients with different stages of CKD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) patients have very low physical function and high rates of cardiovascular disease (CVD) mortality. The objective of the proposed research is to evaluate the effects of dietary supplementation with a pomegranate extract, that contains high amounts of antioxidants, on physical function and CVD risk. Patients with moderate to severe chronic kidney disease that are NOT yet on dialysis tend to have significantly reduced risk factors for cardiovascular disease (and other disorders) compared to dialysis patients. This includes significantly reduced systemic markers of oxidative stress and inflammation. As a result, therapies designed to reduce the risk of CKD co-morbidities may differ significantly in dialysis and pre-dialysis patients. For example, dialysis patients are recommended to INCREASE their intake of dietary protein, while pre-dialysis patients are recommended to DECREASE their protein intake, due to differences in the pathophysiology of the two conditions. The investigators have decided to recruit pre-dialysis patients in addition to dialysis patients in this study because the investigators believe this will help us determine if the efficacy of pomegranate differs between patients with different stages of CKD.

CKD patients will be recruited under 2 phases: CKD patients not receiving dialysis treatment (pre-dialysis patients) will be recruited in the first phase. This will include patients with CKD stage 3-5 that are not yet on dialysis. In the second phase, only CKD patients on dialysis treatment will be recruited. To address these questions, CKD patients will be randomized to the following groups for 12 months: 1) no POM supplementation/control (CON), and 2) oral supplementation with purified pomegranate extract (POM). Patients in the POM group will ingest a 1000 milligram capsule of POM extract, 7 days per week. Patients in the CON group will receive a placebo capsule using the same protocol.

On three occasions, at baseline, 6, and 12 months, each subject will have blood collected to measure plasma markers of oxidative stress (TBARS, lipid peroxides), blood lipid levels, and glucose and insulin levels. Arterial and cardiac structure and function will be measured by vascular ultrasound and echocardiogram, respectively. A 24-hour dietary recall will be used to assess the intake of nutrients. Leg strength will be measured on a resistance exercise machine. Bone density and body composition will be evaluated using dual energy x-ray absorptiometry (DXA). Pre-dialysis subjects will undergo a maximal exercise test to assess their cardiorespiratory fitness level. In dialysis patients, instead of a maximal exercise test, physical function will be measured by a 6-item functional fitness assessment and a 10-meter walk test.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects must be diagnosed with CKD stage 3, 4 or 5 (glomerular filter rate < 59 mL/min).
* 2) Subjects must be ≥ 30 years of age, to increase the probability of having developed significant arterial stiffness.
* 3) Subjects must be willing to be randomized to the control or intervention groups. The health history questionnaire and PAR-Q will be used to determined eligibility.

Subjects must complete a medical history and a nephrologist must sign off on a medical clearance for the subject before they can begin the study.

Exclusion Criteria:

* 1) Subjects < 30 years of age.
* 2) Subjects who are not willing to be randomized to one of the two groups.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Markers of oxidative stress | Circulating markers of oxidative stress will be reduced and serum antioxidant activity will be increased in POM, compared to CON after 12 months of intervention.
Markers of inflammation | Circulating markers of inflammation will be reduced in POM, compared to CON after 12 months of intervention.

SECONDARY OUTCOMES:
Cardiovascular risk | Carotid artery stiffness and CIMT will be reduced in POM compared to CON after 12 months.
Muscular performance | Muscle strength and physical performance will be reduced in CON compared to POM after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wilund, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Champaign-Urbana Dialysis Center, Champaign, Illinois, United States